CLINICAL TRIAL: NCT05874206
Title: Evaluation of Cratos™ Branch Stent Graft System in Treatment of Descending Aorta Lesions
Brief Title: CRATOS - Evaluation of Cratos™ Branch Stent Graft System in Treatment of Descending Aorta Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Endovascular MedTech（Group）Co., Ltd (Industry)
Collaborators: Qmed Consulting A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO_E23-01
Record Dates: First submitted 2023-05-05; First posted 2023-05-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-09

CONDITIONS: Aortic Dissection Type B; Intramural Hematoma; Penetrating Aortic Ulcer
MeSH Terms: conditions — Penetrating Atherosclerotic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TEVAR (Experimental): Thoracic Endovascular Repair (TEVAR) provides a minimally invasive treatment option for descending thoracic aorta (DTA) pathologies.
  Interventions: Device: Cratos™ Stent Graft

INTERVENTIONS:
Device: Cratos™ Stent Graft — Cratos™ Stent Graft TEVAR procedure for the treatment of aortic lesions.

SUMMARY:
The goal of this prospective, interventional, multicentre, single-arm performance objective study is to evaluate efficacy and safety of Cratos™ Branch Stent Graft System in treatment of lesions (dissection, IMH and PAU in descending aorta. The main question[s] it aims to answer are:

* 30-day all-cause Mortality rate
* Composite of the following events from the time of enrolment through 12-month:

  * Device Technical Success
  * Absence of: Aortic rupture, Lesion-related mortality, Disabling Stroke, Permanent paraplegia, Permanent paraparesis, New onset renal failure requiring permanent dialysis, Additional unanticipated post-procedural surgical or interventional procedure related to the device, procedure, or withdrawal of the device system

Participants will come for hospital office visits 1, 6, 12, 24-, 36-, 48- and 60-months post-procedure for the following, but not limited to assessments:

* Physical examination
* Modified Rankin scale
* Tarlov scoring scale
* CTA

ELIGIBILITY:
Inclusion Criteria:

1. Presence of thoracic aortic pathology (Dissection, including IMH and ULP; and PAU) deemed to warrant surgical repair which requires proximal graft placement in Zone 2
2. Age ≥18 years at time of informed consent signature
3. Informed Consent Form (ICF) is signed by Subject or legal representative
4. Must have appropriate proximal aortic landing zone, defined as:

   * Landing zone inner diameters between 23-41 mm
   * The length of landing zone ≥15mm
   * Landing without heavily calcified or heavily thrombosed
   * Dissection Patients: Primary entry tear must be distal to LSA, and proximal extent of the proximal landing zone must not be dissected.
   * For patients with prior replacement of the ascending aorta and/or aortic arch by a surgical graft, there must be at least 2 cm of landing zone proximal to the most distal anastomosis site.
5. Must have appropriate LSA landing zone, defined as:

   * Inner diameters of LSA 5-14 mm
   * Minimum length of Left subclavian artery is 25 mm
   * Target branch vessel landing zone must be in native aorta that cannot be severely tortuous , aneurysmal, dissected, heavily calcified, or heavily thrombosed.
6. Must have appropriate distal aortic landing zone, defined as:

   * Aortic inner diameters between 18-44 mm
   * Landing zone cannot be heavily calcified, or heavily thrombosed.
   * For isolated PAU, outer curvature length must be ≥ 2cm proximal to the celiac artery
   * Landing zone in native aorta

Exclusion Criteria:

1. Concomitant disease of the ascending aorta or aneurysm of the abdominal aorta requiring repair
2. Previous endovascular repair of the ascending aorta
3. Infected aorta, active systemic infection
4. Surgery within 30 days prior to enrolment with the exception of placement of vascular conduit for access .
5. Life expectancy <1 years
6. Myocardial infarction within 6 weeks prior to treatment
7. Stroke within 6 weeks prior to treatment.
8. Pregnant or breastfeeding female
9. Patient has an active systemic infection (e.g., infection requiring treatment with parenteral anti-infective medication) that may place the patient at increased risk of endovascular infection.
10. Degenerative connective tissue disease, e.g., Marfan's or Ehlers-Danlos Syndrome
11. Participation in another drug or medical device study within one year of study enrolment
12. Known history of drug abuse within one year of treatment
13. Tortuous or stenotic iliac and/or femoral arteries preventing introducer sheath insertion and the inability to use a conduit for vascular access
14. Planned coverage of celiac artery
15. Allergic to contrast agents, anaesthetics and delivery materials
16. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
17. Patient with a history of a hypercoagulability disorder and/or is currently in a hypercoagulability state
18. Persistent refractory shock (systolic blood pressure <90 mm Hg)
19. Renal failure defined as patients with an estimated Glomerular Filtration Rate (eGFR) <30 (ml/min/1.73 m2) or currently requiring dialysis
20. Contraindications to antiplatelet drugs and anticoagulants
21. Investigator judged that not suitable for interventional treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30-day
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zimmermann, Prof. Dr., Principal Investigator — Universitätz Spital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided